CLINICAL TRIAL: NCT00705861
Title: A 12 Week, Multi-center, Randomized, Double Blinded, Placebo-controlled, Parallel Group, Fixed Dose Study to Assess the Efficacy and Safety of SK3530 on Erectile Dysfunction in Patients With Diabetes Mellitus
Brief Title: Study to Assess the Efficacy and Safety of SK3530 on Erectile Dysfunction in Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SK3530_DM_III
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Diabetes Mellitus; SK3530
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus | interventions — 2-(5-(4-(2-hydroxyethyl)piperazin-1-ylsulfonyl)-2-n-propoxyphenyl)-5-ethyl-7-n-propyl-3,5-dihydro-4H-pyrrolo(3,2-d)pyrimidin-4-one dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: SK3530

INTERVENTIONS:
Drug: Placebo — Placebo as a substitute of SK3530 100mg
  Arms: 1
Drug: SK3530 — SK3530 100mg
  Other Names: Mvix
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SK3530 on erectile dysfunction in Patients with Diabetes Mellitus.

DETAILED DESCRIPTION:
SK3530 is a potent and selective phosphdiesterase type 5(PDE 5) inhibitor developed for the treatment of erectile dysfunction(ED). Since ED is common in men with Diabetes Mellitus, it is important to determine the efficacy and safety of SK3530 on erectile dysfunction in Patients with Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of type 1 or type 2 diabetes.
* Score below 25 from IIEF EF domain during 4 weeks of treatment run-in period.
* Failure rate above 50% from sexual attempt above 4 during 4 weeks of treatment run-in period.

Exclusion Criteria:

* Lab abnormality.
* Uncontrolled diabetic mellitus(HbA1c > 12%).
* High or low blood pressure, orthostatic hypotension.
* Hyper- or hypo-thyroidism.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Erectile Function domain score (sum of Question 1,2,3,4,5 and 15) of the International Index of Erectile Function (IIEF) Questionnaire | 0, 4, 8, 12week

SECONDARY OUTCOMES:
the score from : 1) IIEF Q3 & Q4, 2) other domains of IIEF, 3) Sexual Encounter Profile(SEP)Q2 and Q3, 4) Life Satisfaction Checklist, 5) Global Efficacy Assessment Question(GEAQ) | 0, 4, 8, 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Chul Park, MD, PhD, Principal Investigator — BNUH
Locations (1):
- SK Chemicals Co., Ltd, Seoul, South Korea